CLINICAL TRIAL: NCT06718478
Title: First in Human Study of SakuraBead for Genicular Artery Embolization to Treat Pain Secondary to Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CrannMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI520
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis (OA) of the Knee; Osteoarthritis Knee Pain; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis; Osteoarthritis
Keywords: Genicular Artery Embolization; GAE; Knee Embolization; Knee OA; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genicular Artery Embolization (GAE) (Experimental): Temporary Embolization of Genicular Arteries using SakuraBead Resorbable Microspheres
  Interventions: Device: SakuraBead Resorbable Microspheres

INTERVENTIONS:
Device: SakuraBead Resorbable Microspheres — Temporary Embolization of Genicular Arteries using SakuraBead Resorbable Microspheres

SUMMARY:
A prospective, single-centre, single-arm, unmasked, First in Human study that aims to evaluate the safety and efficacy of SakuraBead resorbable microspheres in adult patients suffering from pain secondary to knee osteoarthritis.

DETAILED DESCRIPTION:
To evaluate safety and efficacy of SakuraBead for the treatment of pain secondary to knee osteoarthritis. Treatment will be performed on up to 15 patients who will be followed up for a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able and willing to provide written informed consent, and
2. Clinical diagnosis of knee OA, and
3. Moderate to severe knee pain (VAS ≥ 5), and
4. Pain refractory to at least 3 months* of conservative therapies (anti-inflammatory drugs, or physical therapy, or muscle strengthening, or intra-articular injections), and
5. Kellgren-Lawrence grade 1, 2 or 3 on radiograph of the knee, and
6. Age 40 years or older.
7. Subject has confirmed evidence of knee OA, defined as an angiographic 'blush' pattern (radiographic) in one or more of the target genicular artery(ies).

Exclusion Criteria:

1. Severe knee OA (Kellgren-Lawrence grade 4)
2. Current infection of target joint, or
3. Life expectancy less than 24 months, or
4. Known advanced atherosclerosis as defined by history of lower extremity or pelvis arterial bypass graft, lower extremity or pelvis arterial stent placement or prior history of vascular claudication, or
5. Rheumatoid or known serologic diagnosis of autoimmune arthritis, or
6. Prior knee replacement surgery in the target knee, or
7. Complete meniscal or cruciate tear that requires surgery, or
8. History of uncorrectable coagulopathy, or
9. Prior iodinated contrast reaction resulting in anaphylaxis, or
10. Pregnant and/or lactating female, or
11. At the discretion of the Principal Investigator
12. Subject has evidence of arterial occlusion precluding catheterization.
13. Subject has occlusion of the genicular arteries.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Decrease of pain on Visual Analogue Scale (VAS) at 1 month follow-up. | 1 month
Genicular Artery Embolization (GAE) without a major device- or procedure-related complication at 1 month follow-up | 1 month

SECONDARY OUTCOMES:
Reduction in global Western Ontario and McMaster University Osteoarthritis Index (WOMAC) questionnaire at 1 month, 3 months and 6 months follow-up | 1, 3 and 6 months
Reduction of previously initiated OsteoArthritis (OA) medical therapy at 3- and 6-months follow-up | 3 and 6 months
Decrease of pain on Visual Analogue Scale (VAS) at 3 and 6 months | 3 and 6 months
No major device- or procedure-related complication at 3 and 6 months | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Republican Specialized Scientific and Practical Medical Center of Therapy and Medical Rehabilitation, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No